CLINICAL TRIAL: NCT04995146
Title: Implementing International Standards of Practice in A Low Resource Country by Blended Training Modules to Improve Stroke Care
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Other Study IDs: FUI/CTR/2020/8
Record Dates: First submitted 2021-02-13; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective 3 months cohort (admitted stroke patients)
  Interventions: Other: Clinical stroke extended management pathway
- Prospective pre-implementation "standard of core care quality measures" cohort
  Interventions: Other: Clinical stroke extended management pathway
- Prospective post-implementation "standard of core care quality measures" cohort
  Interventions: Other: Clinical stroke extended management pathway

INTERVENTIONS:
Other: Clinical stroke extended management pathway — 1. Extracranial imaging
  2. ECG in 2-7 days
  3. DVT prophylaxis
  4. Stroke educational material for patient and family Removal of Foley's catheter and start bladder management
  5. Discharged on: Antithrombotic therapy OR Anticoagulation therapy▸ Antihypertensives ▸ Statins/cholesterol lower agent ▸ Antidiabetic agent
  6. Fasting lipid profile, HbA1c
  7. Holter monitor
  8. Specialized workup for young stroke
  9. PFO Study, MES Study
  10. Referral to: ▸ Rehabilitation specialist ▸ Speech therapist ▸ Dietician ▸ Occupational therapist ▸ Medical team
  11. Follow-up: CTA, CT angiography; HbA1c, glycated haemoglobin; MRA, MR angiography
  12. Follow-up plan and 90 day mRS

SUMMARY:
Lack of proper stroke care delivery leads to poor patient outcomes in middle- and low-income countries that can be improved by implementation of international standards. We aim to determine feasibility of implementing stroke core measures and training through blended learning modules in resource poor countries to improve stroke outcomes.

DETAILED DESCRIPTION:
Background: Lack of proper stroke care delivery leads to poor patient outcomes in middle- and low-income countries that can be improved by implementation of international standards. We aim to determine feasibility of implementing stroke core measures and training through blended learning modules in resource poor countries to improve stroke outcomes.

Methods: The project will be conducted across four hospitals in Pakistan in three phases. First stage will include retrospective collection of data for the preceding 4 weeks from start. In stage II, 3 months data will be collected before implementation of core measures. The stepwise training of staff will begin simultaneously, and data will continue to be collected. In stage III by the end of 3 months of stage II, core measures will be implemented as standard of care and patients will be enrolled for another 3 months. Outcomes measures will be successful implementation of the stroke care model as measured by survey done at the end and patient outcomes including in-hospital complication rates, length of hospital stay, patient and caregiver education, mRS at 3 months after discharge, post discharge complications and re-stroke rate. Data will be compared against published data from Pakistan and between patients in the first and last 3 months of the project. Statistical analyses will include appropriate mixed-effects multivariate regression models (i.e., linear and logistic) to model the relationship between clinical measures and patient safety. Degree of correlation across each symptom predictor will be measured. This study will not involve thrombolytic therapy or thrombectomy. However, the study will not provide any hindrance to implementation of such therapy and will not include such patients in analysis.

Discussion: At least one third of stroke survivors in Pakistan die due to recurrent vascular events and complications of stroke in absence of core measures. Prevention practices and stroke care are significantly underutilized in low- and middle-income countries but can be improved most efficiently by improving care delivering process without additional burden on resources by following American Heart Association "Get With The Guidelines" Stroke (GWTG-Stroke) program, Royal College of Physicians UK and European Guidelines, regardless of thrombolysis or thrombectomy. This feasibility study aims to develop a multidisciplinary comprehensive stroke team model with gradual integration of staff training, nursing care, therapy and patient education.

ELIGIBILITY:
Inclusion Criteria:

Acute onset of Symptoms in the last 24 hours suggestive of stroke Age > 18 years Ischemic or hemorrhagic stroke

-

Exclusion Criteria:

Presenting after 24 hours of onset of symptoms Alternate explanation for presenting symptoms (stroke mimics) Family (Surrogate Decision Maker) or next of kin/ patient refusal for participation Transfer of care from another department or hospital Care needed in another department (e.g, ICU, other department) GCS (Glasgow Coma Scale) below 5 or End of life care initiated TIA (Transient Ischemic Attack)

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute stroke symptoms as deemed by treating physicians presenting to the ED will be enrolled. Normative data from the general population will be used where needed for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Post Core Measure Delivery | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
  • Primary outcome measure will be successful implementation of the stroke care model as measured by survey done at the end assessing engagement and ability to continue the program in future and ability to implement the program across institutions. This will be measured by the NIHSS training, stroke education, awareness of core measures, the regularity of following the core measure and data collection.

SECONDARY OUTCOMES:
Modified Rankin Scale | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 days
  Modified Rankin Scale is a 6 point disability scale from 0-6, and a greater score means worse outcome.
New ischemic stroke or Transient Ischemic Attack: | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 days
Hemorrhagic transformation: | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 days
Intracranial hemorrhage: | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 days
Death | From date of inclusion in the study until the date of discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No